CLINICAL TRIAL: NCT05551442
Title: Xu Pu, Director, Clinical Researcher
Brief Title: A Controlled Study of Improved Javelin Side Recumbent Position and Conventional Postural Placement
Status: Completed | Type: Observational
Sponsor: Guiyang Maternal and Child Health Care Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Xu Pu
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2021-12

CONDITIONS: Nurse-Patient Relations
Keywords: ureteropelvic junction obstruction
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- In control group A,: In control group A, we adopted the conventional lateral position
  Interventions: Procedure: To explore the comparative study of different positioning methods in robot assisted laparoscopic pyeloplasty.; Device: To discuss the comparative study of different position placement methods of renal pelvis ureteroplasty on the Da Vinci robotic Xi platform
- control group B: control group B adopted the lumbar bridge cushion lateral position
  Interventions: Procedure: To explore the comparative study of different positioning methods in robot assisted laparoscopic pyeloplasty.; Device: To discuss the comparative study of different position placement methods of renal pelvis ureteroplasty on the Da Vinci robotic Xi platform
- observation group C: observation group C adopted the modified javelin lateral position
  Interventions: Procedure: To explore the comparative study of different positioning methods in robot assisted laparoscopic pyeloplasty.; Device: To discuss the comparative study of different position placement methods of renal pelvis ureteroplasty on the Da Vinci robotic Xi platform

INTERVENTIONS:
Procedure: To explore the comparative study of different positioning methods in robot assisted laparoscopic pyeloplasty. — The incidence of surgical positioning time and secondary berths, surgical time, intraoperative blood loss and intraoperative complications were compared among the three groups.
Device: To discuss the comparative study of different position placement methods of renal pelvis ureteroplasty on the Da Vinci robotic Xi platform — To discuss the comparative study of different position placement methods of renal pelvis ureteroplasty on the Da Vinci robotic Xi platform

SUMMARY:
The Da Vinci surgical robot Xi system assisted laparoscopic pyeloureteroplasty uses the improved javelin side lying position, which can alleviate the unsafe factors of falling from the bed caused by the conventional posture, shorten the time of placing the posture5, prevent the possible pressure injuries and intraoperative complications caused by the conventional posture surgery, and the operation is more simple and convenient. The mechanical arm of the Da Vinci robot will not have the potential risk factors of crushing the head, face and trunk of the patient during the entire operation process, It is safe and reliable, making the whole process of positioning convenient and time-saving. It can not only improve the connection efficiency of each operation, but also ease the work intensity of nurses and reduce the incidence of robot secondary berths. Operator satisfaction. It is safe and reliable to achieve good results, improve the operation safety, effectively avoid intraoperative and postoperative complications, and ensure the operation safety of patients, which is worth promoting.

DETAILED DESCRIPTION:
To discuss the comparative study of different localization methods in robot-assisted laparoscopic epirenoplasty.

From December 2021 to January 2022, the researchers selected 60 participants to undergo laparoscopic pyroplasty assisted by the Da Vinci Robotic Xi system. Depending on the order of the surgeries, the researchers randomly assigned them， the subjects into three groups: control group A, control group B and observation group C, each with 20 cases. In control group A, we adopted the conventional lateral position, control group B adopted the lumbar bridge cushion lateral position, and observation group C adopted the modified javelin lateral position, The operation time, secondary berth incidence, operation time, intraoperative blood loss and the incidence of intraoperative complications were compared among the three groups.

ELIGIBILITY:
Selection Criteria:

1. Clinical diagnosis of obstruction at the renal pelvis ureteral junction.
2. Must be able to fit the treatment done under the robot platform

Exclusion Criteria:

1. Patients who can use balloon dilation to achieve the therapeutic purpose
2. Open surgery is required

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: From December 2021 to January 2022, 60 patients with da Vinci robotic Xi system assisted laparoscopic pyelonegal ureteroplasty surgery were selected in our hospital, and according to the order of surgery, we randomly divided the study objects into three groups, namely control group A, control group B and observation group C 20 cases each, control group A We took the conventional lateral lying position, control group B adopted the lumbar bridge pad high lateral recumbent position, observation group C adopted the design to improve the javelin side lying position, compared the three groups of surgical positioning time, secondary berth incidence, and surgical time 3. Intraoperative blood loss and incidence of intraoperative complications.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-01-09 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
The da Vinci surgical robot Xi system assists laparoscopic pyeloneuroplasty with an absolute advantage in the modified javelin lateral recumbent position | From December 2021 to January 2022
  The use of modified javelin side recumbent position during surgery can alleviate the unsafe factors of falling from the bed caused by conventional positioning, which is safe and reliable, and achieves good results

CONTACTS AND LOCATIONS:
Overall Officials: Jing P Liu, doctorat, Study Director — Guizhou Provincial People's Hospital
Locations (1):
- GuiyangMaternalChildHCH, Guiyang, China

IPD SHARING:
Plan to Share IPD: Yes
A study design of the modified lateral position of javelin and the conventional position of body in the operation of pediatric ureteropelvic junction obstruction with Da Vinci Xi platform
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code